CLINICAL TRIAL: NCT06802926
Title: A Single Center Pilot Trial of Preliminary Effect of Colchicine on Graft Failure in Patients Underwent CABG
Brief Title: Pilot Trial of Colchicine for Graft Failure in CABG
Acronym: CoCAB-Pilot
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhu yunpeng, Professor and Director of Clinical Research, Department of Cardiovascular Surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2025-777
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: CABG; Graft Failure; Colchicine
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Oral Colchicine 0.5mg qd for 1 year
  Interventions: Drug: Colchicine
- Blank control (No Intervention): No Oral Colchicine therapy

INTERVENTIONS:
Drug: Colchicine — Oral Colchicine 0.5mg qd for 1 year
  Arms: Colchicine

SUMMARY:
The goal of this pilot trial is to to evaluate the preliminary effect of oral colchicine therapy on graft outcomes in patients underwent primary isolated CABG.

The main questions it aims to answer is:

1. Whether the oral colchicine therapy may reduce the failure outcome of grafts after CABG.
2. Whether it is feasible to construct a muticenter powered trial to test the superiority hypothesis.

Researchers will compare colchicine to none to see if colchicine works.

Participants will

1. Take oral colchicine (0.5mg daily) therapy for 12 months after CABG.
2. Clinical follow-up at Month 1, 6, and 12 after CABG.
3. Protocol-driven CCTA at Week 1 and Month 12 after CABG.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old，
* Any sex，
* Signed informed consent，
* Within 3 days after a successful isolated CABG

Exclusion Criteria:

* Allergy,
* Hematopoietic dysfunction,
* Moderate to severe hepatic dysfunction,
* Moderate to severe renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The Graft Failure Rate at 1 year | at 1 year post-CABG
  A protocol-driven CCTA will be used to evaluate the graft outcome at 1 year after CABG. Fitzgibbon Grade B/S/O is definned as graft failure.

SECONDARY OUTCOMES:
The time to first 5-point Major Adverse Cardiovascular Event (MACE-5) | within 1 year post-CABG
  MACE-5 is a composite of all-cause death, myocardial infarction, stroke, unplanned revascularization, and rehospitalization due to unstable angina.
The rate of new perioperative atrial fibrillationat (PAF) within 1 week after CABG | within 7 days post-CABG
  PAF will be detected through continuous electrocardiographic monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Study Chair — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China; Yunpeng Zhu, MD, Principal Investigator — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR